CLINICAL TRIAL: NCT02493582
Title: The Randomized, Controlled Clinical Trial of Apatinib Plus CIK as the Third Line Therapy for Lung Adenocarcinoma Patients With Wild-Type EGFR
Brief Title: The Study of Apatinib Plus CIK as the Third Line Therapy for Advanced Lung Adenocarcinoma Patients With Wild-Type EGFR
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First People's Hospital of Changzhou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAA
Record Dates: First submitted 2015-07-07; First posted 2015-07-09 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-02

CONDITIONS: Adenocarcinoma of Lung
Keywords: CIK; Apatinib; Lung Adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma of Lung | interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Apatinib alone (Other): Apatinib(YN968D1) ,850mg,p.o.,qd,continuous.
  Interventions: Drug: Apatinib
- Apatinib+CIK (Experimental): Apatinib(YN968D1) ,850mg,p.o.,qd,continuous. plus autologous cytokine-induced killer cells 3 cycles,every 1 year,continuous.
  Interventions: Biological: Cytokine-Induced Killer Cells; Drug: Apatinib

INTERVENTIONS:
Biological: Cytokine-Induced Killer Cells — CIKs are used with Apatinib to treat lung adenocarcinoma patients with wild-type EGFR
  Other Names: CIK
  Arms: Apatinib+CIK
Drug: Apatinib — Advanced lung adenocarcinoma patients with wild-type EGFR take Apatinib 850mg qd by mouth.
  Other Names: YN968D1

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of Apatinib combined with cytokine-induced killer cell (CIK) vs Apatinib alone as the third line therapy for advanced lung adenocarcinoma patients with wild-type EGFR

DETAILED DESCRIPTION:
400 patients with stage IIIB & IV lung adenocarcinoma who had received surgery and chemotherapy,will be randomly divided into group A（Apatinib plus CIK treatment ) or group B（Apatinib), and the randomize ratio will be 1:1. Patients in group A will receive 3 cycles of CIK treatment (every 1 year) and Apatinib (continuous).Patients in group B will receive only Apatinib (continuous) .

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed Lung adenocarcinoma
* Wld-type EGFR
* Stage IIIB/IV
* Failure to prior chemotherapy
* Life expectancy of more than 3 months
* Tissue sample desired for genomic study
* Age ≥ 18 years
* Performance status (WHO) < 3
* Adequate bone marrow function (absolute neutrophil count>1000/mm^3, platelet count > 100000/mm^3, hemoglobin > 9gr/mm^3)
* Adequate liver (bilirubin < 1.5 times upper limit of normal and SGOT/SGPT < 2 times upper limit of normal) and renal function (creatinine < 2mg/dl)
* Presence of two-dimensional measurable disease. The measurable disease should not have been irradiated
* Informed consent

Exclusion Criteria:

* Lung squamous cell carcinoma or other types of Non-Small cell lung cancer
* Small cell lung cancer
* Have previously received TKIs
* Hemoglobin<8.0 g/dL,White blood cell <3 X 10^9/L;Platelet count <75 X 10^9/L; alanine aminotransferase, glutamic-oxalacetic transaminase, blood urine nitrogen and creatinine more than normal limits on 3.0 times
* Known or suspected allergy to the investigational agent or any agent given in association with this trial
* Pregnant or lactating patients
* Known history of Human Immunodeficiency Virus (HIV), Hepatitis C Virus (HCV) or TreponemaPallidun (TP) infection
* Patients who are suffering from serious autoimmune disease
* Patients who had used long time or are using immunosuppressant
* Patients who had active infection
* Patients who are suffering from serious organ dysfunction
* Patients who are suffering from other cancer
* Other situations that the researchers considered unsuitable for this study.
* Other concurrent uncontrolled illness

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2015-07; Primary Completion 2030-07 (Estimated); Study Completion 2033-07 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | 3 months

SECONDARY OUTCOMES:
Progression-Free-Survival (PFS) | 3 months

OTHER OUTCOMES:
Number of participants with Adverse events | 1 month